CLINICAL TRIAL: NCT00255931
Title: Biobehavioral Intervention in Heart Failure
Brief Title: Impact of a Psychological Biofeedback-Relaxation Intervention on Clinical, Physical and Psychological Outcomes in Patients With Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Debra Moser, Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8567; R01NR008567 (NIH); R01NR008567-01A1 (NIH)
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; Biofeedback-Relaxation; Cognitive Behavioral Therapy
MeSH Terms: conditions — Heart Failure | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (Placebo Comparator)
  Interventions: Behavioral: Attention Placebo
- 3 (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy and Relaxation/biofeedback
  Arms: 1
Behavioral: Attention Placebo — Untrained relaxation
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of biofeedback-relaxation combined with cognitive behavioral therapy on clinical, physical and psychological outcomes in patients with heart failure.

DETAILED DESCRIPTION:
The long-term aim of this program of research is to improve physical and psychological health outcomes of adults with heart failure (HF). The specific aims of the randomized, controlled clinical trial are to test the effects of biofeedback-relaxation therapy in HF patients on rehospitalizations, cardiac mortality and quality of life, and on the secondary end-points of perceived control, anxiety, depression, skin temperature, plasma norepinephrine levels, and heart rate variability (HRV).

In the 1990s, HF emerged as a significant public health threat and reached epidemic proportions. Heart failure incidence and prevalence are expected to increase worldwide, and its impact to worsen dramatically. Individuals with HF suffer incapacitating physical symptoms, emotional distress, impaired quality of life, repeated rehospitalizations, and premature death. To combat the rising HF epidemic, it is crucial that researchers study new strategies to improve outcomes. Despite its potential as an effective partner to drug therapy, the role of nonpharmacologic intervention in HF management has received relatively little attention.

One may argue that drug therapy is effective enough that resources need not be expended on research of nonpharmacologic therapies. However, three points argue against this stance. First, despite substantial advances made in HF treatment with drug therapy, morbidity and mortality remain unacceptably high. As Kannel states, "innovations in treatment of...HF have thus far made a disappointingly small improvement in its…outlook". Second, although drug therapy frequently provides significant improvement in symptoms and functional ability, quality of life may not improve. This outcome is important for patients with HF because poorer quality of life independently predicts morbidity and mortality. Third, nonpharmacologic strategies can have effect sizes for important HF outcomes (e.g., rehospitalization rates/mortality and quality of life) that are similar to those seen with drug therapy. Recent studies demonstrated these therapies substantially improve outcomes beyond the level seen in the same patients with pharmacologic therapy.

Biofeedback-relaxation therapy is an innovative and promising nonpharmacologic strategy. An optimally effective treatment should have a beneficial effect on both pathophysiological and psychological manifestations of the target condition. This goal is especially important for a condition like HF, which has a profoundly negative impact on physical and psychological function. Hallmark pathophysiology in HF includes intense neurohumoral activation, initiated and sustained by the sympathetic nervous system (SNS), with marked vasoconstriction. Adverse psychological manifestations of chronic HF include feelings of loss of control, anxiety and depression. Both neurohumoral activation and the psychological consequences of HF contribute to poor quality of life, frequent HF hospitalizations, and increased mortality. As shown in the model in Figure 1, biofeedback-relaxation therapy takes three complementary, but separate pathways to improve outcomes. This biobehavioral therapy decreases SNS activation (as reflected by HRV and plasma norepinephrine), produces stress reduction (as reflected by changes in perceived control, anxiety and depression), and results in vasodilation (as reflected by skin temperature). Biofeedback-relaxation therapy can have a powerful influence because of these separate, yet complementary effects. For example, SNS activation is directly decreased by biofeedback-relaxation therapy, but also indirectly as a result of stress reduction with increased control, and decreased anxiety and depression. As a result of its physical and psychological effects, biofeedback-relaxation could have a clinically meaningful impact on rehospitalizations, survival and quality of life. For these reasons, biofeedback-relaxation may be an effective adjunct to pharmacologic therapy in the management of HF. Thus, the purpose of the proposed research is to examine the impact of biofeedback-relaxation training on HF patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of chronic advanced HF. Other sample selection criteria include: 1) on stable doses of HF medication for at least one month; and 2) not referred for heart transplantation.

Exclusion Criteria:

* Patients will be excluded if they have: 1) valvular heart disease (as a primary cause of their HF; can have it if the primary cause is ischemic, hypertensive or idiopathic), peripartum heart failure, myocarditis; 2) history of cerebral vascular accident (CVA) within previous 3 months or major stroke sequelae; 3) history of major extremity vascular problems; 4) recent (within 3 months) myocardial infarction (MI); 5) coexisting terminal illness; 6) systolic blood pressure less than 80 mmHg; or 7) previous experience with biofeedback, relaxation .

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2004-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Examination of the impact of biofeedback-relaxation training on HF patient outcomes. | Baseline, 3-, and 12-Months

SECONDARY OUTCOMES:
Perceived Control | Baseline, 3-, and 12-Months
Anxiety | Baseline, 3-, and 12-Months
Depression | Baseline, 3-, and 12-Months
Skin Temperature | Baseline, 3-, and 12-Months
Heart Rate Variability | Baseline, 3-, and 12-Months
Plasma Norepinephrine | Baseline, 3-, and 12-Months

CONTACTS AND LOCATIONS:
Overall Officials: Debra Moser, DNSc, RN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States